CLINICAL TRIAL: NCT01642329
Title: Portuguese Registry on Acute Coronary Syndromes
Acronym: ProACS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Portuguese Society of Cardiology (Other)
Responsible Party: Sponsor
Other Study IDs: ProACS; ProACS (Registry Identifier: Portuguese Registry on Acute Coronary Syndromes)
Record Dates: First submitted 2012-07-13; First posted 2012-07-17 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-10

CONDITIONS: Acute Coronary Syndrome
Keywords: Myocardial Infarction; Angina, Unstable
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction; Angina, Unstable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — no samples retained
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this Registry is creating a database management that allows continuous monitoring characteristics, evolution, prognostic indicators and management of patients with ACS admitted in Portuguese Hospitals, and identify the appropriateness of clinical practice recommendations for diagnosis and treatment of ACS and monitor its evolution.

DETAILED DESCRIPTION:
Cardiovascular diseases remain the principal causes of death in Portugal and approximately one quarter of these are directly to ischemic heart disease, especially Acute Coronary Syndromes (ACS).

In order to reduce mortality for ACS, a significant number of new drugs and new techniques have been introduced into clinical practice, resulting in important heterogeneity of approach and treatment of patients with ACS.

The Portuguese Society of Cardiology have sought to review and incorporate in its recommendations the evidence to date, with the aim to standardize diagnosis and treatment of patients with ACS, which is not always able to in daily practice.

Since it is essential to characterize the national reality of the ACS, the Portuguese Society of Cardiology has promoted the Portuguese registry on Acute Coronary Syndromes, aimed at bridging the knowledge gaps in this area of cardiovascular disease.

This will include all adult patients (≥ 18 years) diagnosed with Acute Coronary Syndrome (ACS) with <48 hours of evolution. The inclusion is of responsibility of the last service of Cardiology where the patient was hospitalized. The ACS is set to the presence of angina at rest last 48 hours, with 1) ischemic electrocardiographic changes ST-segment deviations or negative T waves, and / or 2) elevation of biomarker (cardiac troponin and CK-MB) above the reference value. For diagnosis ACS with ST elevation is considered to be persistently elevated (> 30 minutes) of the ST segment. The rest should be considered as ACS ST-segment elevation. In the absence of angina, the SCA will be considered consistent elevation (curve ascending / descending) biomarker (above reference value for cardiac troponin or higher 2 times the value of reference to the CK-MB) associated with other clinical manifestations such as ill-defined chest discomfort or dyspnea.

Are included patients participating in clinical trials

Are excluded patients with MI after revascularization procedures (EAM type 4 and 5) and MI type 2 (classification according to the redefinition of Myocardial Infarction, 2007 the Joint ESC / ACCF / AHA / WHF Task Force)

ELIGIBILITY:
Inclusion Criteria:

* presence of angina at rest last 48 hours, with: 1) ischemic electrocardiographic changes - ST-segment deviations or negative T waves, and / or 2) elevation of biomarker(cardiac troponin and CK-MB) above the reference value.

Exclusion Criteria:

* patients with MI after revascularization procedures (EAM type 4 and 5) and MI type 2 (classification according to the redefinition of Myocardial Infarction, 2007 the Joint ESC / ACCF / AHA / WHF Task Force).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients with Acute Coronary Syndrome (ACS) with <48 hours of evolution, admitted to Portuguese Hospitals.
Sampling Method: Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2002-01; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Hospital mortality in patients admitted for acute coronary syndrome | Hospital dead in patients admitted with acute coronary syndrome
  Evaluation of hospital mortality rate of patients admitted for acute coronary syndrome

SECONDARY OUTCOMES:
major adverse cardiac events (MACE) | In-hospital MACE in patients admitted for acute coronary syndrome
  MACE In-hospital major adverse cardiac event (death, myocardial infarction,heart failure,stroke,)

OTHER OUTCOMES:
Major bleeding | In hospital major bleeding
  In Hospital major bleeding based on GUSTO definition

CONTACTS AND LOCATIONS:
Overall Officials: Jorge V Mimoso, MD, Principal Investigator — Portuguese Society of Cardiology
Locations (1):
- CNCDC, Coimbra, Coimbra District, Portugal

REFERENCES:
- See also: Portuguese Society of Cardiology — http://www.spc.pt/spc/